CLINICAL TRIAL: NCT05734963
Title: ORganoid GeneratioN Study for Cancer
Acronym: ORIGINS
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5396
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with histologically confirmed cancer
  Tissue, blood and saliva samples collected before and after surgery and before and after any adjuvant therapy. Molecular profiling, DNA sequencing, gene expression analysis
  Interventions: Genetic: DNA sequencing, RNA gene expression analysis, molecular profiling

INTERVENTIONS:
Genetic: DNA sequencing, RNA gene expression analysis, molecular profiling — Growth of organoids from tissue samples, collection of tissue, blood and saliva samples for DNA sequencing, RNA gene expression analysis, molecular profiling

SUMMARY:
ORIGINS - a multi-site sample collection study to establish patient-derived pre-clinical models for cancers

DETAILED DESCRIPTION:
People who develop cancer can often be cured if they are suitable for surgery or radiotherapy. However, a proportion of these cancers return, at which point the available treatment options are often not very effective. Our understanding of the biology of many cancers is limited, and we don't understand why some cancers are cured by surgery or radiotherapy and some are not. A better understanding of the biology of cancers could help develop new treatments, or improvements to current treatments, and this might increase the number of patients who can be cured of their disease.

One way to improve the understanding we have of the biology is to look in detail at cancer samples taken from the from patients. The problem with this is that often samples are small, and the tumour tissue sample itself already dead once removed from where it was growing, which can limit the analyses that are possible. A potential solution for this is to take cancer tissue from patients and try to directly grow the cells in the laboratory. Keeping the cancer cells alive in the laboratory can be difficult but has been shown to be possible in a number of different types of cancer. This kind of model is sometimes known as an "organoid". If successfully established, it means more tests can be done to find out how the cancer is working.

This study is looking at collecting samples of a person's cancer to see if we can develop these models from patients being treated for different cancers. We will ask people who are having surgery for cancer whether we can take samples from their tumour to try and achieve this. Some additional blood tests will be taken alongside the usual blood tests before and after surgery, without an additional blood draw, and before and again after any adjuvant therapy is completed. A collection of saliva will also be requested at these times and we will ask people whether they are happy for us to collect any previous tissue samples, or nay that are subsequently collected when they are being followed up, to allow comparison with the samples collected as part of this study.

The main goal of this study is to see if organoids can be established in our laboratories. If these models are successfully established, we will compare them to the original tumour to check they are a good match biologically. After this we can use them to understand how the cancer works and try out new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with histologically proven or suspected cancer undergoing an interventional procedure, such as surgery or biopsy
* Ability to give informed consent for biological sample collection

Exclusion Criteria:

* Unable to undergo sample collection
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven or suspected cancer undergoing an interventional procedure, such as surgery or biopsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2031-04-12 (Estimated); Study Completion 2031-04-12 (Estimated)

PRIMARY OUTCOMES:
Establish patient-derived organoid (PDO) model for cancers | Time Frame: Through study completion, expected duration of 9 years
  Establish patient-derived organoid (PDO) model for cancers

SECONDARY OUTCOMES:
To collection contemporaneous biological samples from patients with cancer before and after surgery/biopsy, and again after any adjuvant therapy | Time Frame: Through study completion, expected duration of 9 years
  To collection contemporaneous biological samples from patients with cancer before and after surgery/biopsy, and again after any adjuvant therapy - including blood, saliva and tissue, for molecular profiling, including extraction of DNA for sequencing, RNA
To collect tumour tissue to facilitate evolutionary analysis with molecular analysis of multiple regions | Time Frame: Through study completion, expected duration of 9 years
  To collect tumour tissue to facilitate evolutionary analysis with molecular analysis of multiple regions
Retrieval and analysis of archival primary tissue blocks for comparison where available | Time Frame: Through study completion, expected duration of 9 years
  Retrieval and analysis of archival primary tissue blocks for comparison where available
To establish co-culture tumour/stroma/immune cell models | Time Frame: Through study completion, expected duration of 9 years
  To establish co-culture tumour/stroma/immune cell models
To observe associations between molecular and clinicopathological data | Time Frame: Through study completion, expected duration of 9 years
  To observe associations between molecular and clinicopathological data

CONTACTS AND LOCATIONS:
Overall Officials: Ben O'Leary, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No